CLINICAL TRIAL: NCT05427773
Title: (In)Voluntary Assessed Quadriceps Muscle Endurance in Patients With Chronic Obstructive Pulmonary Disease: a Cross-sectional Observation Study.
Brief Title: (In)Voluntary Assessed Quadriceps Muscle Endurance in COPD
Acronym: Bionic
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1132321
Record Dates: First submitted 2022-06-13; First posted 2022-06-22 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Peripheral muscle endurance; Electrical stimulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective is to assess the relation between involuntary and voluntary assessed quadriceps muscle endurance in patients with COPD. We hypothesized a good correlation (>0.8) between the measurements.

DETAILED DESCRIPTION:
Rationale: Quadriceps muscle endurance is reduced in patients with COPD. However, no consensus has been reached yet on the best method to evaluate quadriceps muscle endurance. One important aspect is the large variety in protocols and devices used around the world. Commonly used and reliable measures are voluntary protocols performed on a computerized dynamometer. However, these voluntary measurements might also be influenced by external factors as patients effort or motivation. Therefore, it is important to evaluate the relation between voluntary and involuntary (i.e. electrical stimulated) assessed quadriceps muscle endurance.

Objective(s): The primary objective is to assess the relation between involuntary and voluntary assessed quadriceps muscle endurance in patients with COPD.

Study design: Cross-sectional observation study.

Study population: 20 COPD patients who perform baseline assessment at the pulmonary rehabilitation centre at Radboudumc (Nijmegen, the Netherlands).

Intervention: not applicable

Main study parameters/endpoints: The primary outcome will be the electrically evoked isometric quadriceps muscle endurance (fatigue resistance) and voluntary isokinetic (work fatigue index5) and isometric quadriceps endurance (time).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: BURDEN: All measurements are part of standard care, except for one questionnaire and (involuntary) electrical assessed quadriceps function. Thus, the additional burden for the patient is one additional measurement of approximately 70 minutes. RISKS: Performance of electrically evoked assessment of muscle function is not associated with a health risk. This procedure is non-invasive and not painful and performed routinely at the department of Physiology (Radboudumc, Nijmegen). Therefore, no safety risk is involved.

BENEFIT: The benefits will be high as it will provide more insight in the relation between voluntary and involuntary assessed quadriceps muscle endurance. This insight is necessary to optimize the clinical assessment of muscle endurance in patients with COPD.

GROUP RELATEDNESS: This will be the first study in which the relation between voluntary and involuntary assessed quadriceps muscle endurance in COPD will be investigated. These results will also be valuable for other diseases/conditions in which isolated muscle endurance should be assessed like asthma, pulmonary hypertension, etc.

ELIGIBILITY:
Inclusion Criteria:

* COPD, based on GOLD classification
* Clinically stable according to the pulmonary physician, i.e. no exacerbation and/or hospitalization within the previous 4 weeks
* Age between 40-80 years
* Take part in the pulmonary rehabilitation program at Radboudumc (Nijmegen)

Exclusion Criteria:

* Inability to understand the Dutch language
* Musculoskeletal and neurological problems influencing quadriceps muscle function testing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD that start with the pulmonary rehabilitation program at the Radboudumc in Nijmegen.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Electrically evoked fatigue resistance (%) | Performed in first week of pulmonary rehabilitation program
  Fatigue resistance (%) is the decline in muscle force generated using electrical stimulation.
Voluntary isometric quadriceps endurance (time to fatigue). | Performed in first week of pulmonary rehabilitation program
  Voluntary isometric quadriceps endurance (time to fatigue in seconds) is determined on the computerized dynamometer. The isometric endurance test protocol is performed by asking participants to maintain, for as long as possible, an isometric quadriceps contraction representing 60% of the individual isometric maximal voluntary contraction (MVC) force. The test will be ended if the force of the contraction was less than 50% of the MVC for three consecutive seconds.
Voluntary isokinetic work fatigue index. | Performed in first week of pulmonary rehabilitation program
  Voluntary isokinetic work fatigue (%) is the decline in work over 30 repetitions determined on the computerized dynamometer. The isokinetic protocol consists of 30 contractions at an angular velocity of 90°/s with maximal effort during extension and passive (submaximal) flexion.
  Work fatigue index = *work first 5 repetitions - work last 5 repetitions) / work first 5 repetitions * 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands